CLINICAL TRIAL: NCT03188900
Title: New Therapeutic Strategy Against Preeclampsia: Angiogenic Switch to Physiological State by Extracorporeal Removal of sFlt-1
Brief Title: Blood Collection to Validated New Therapeutics Strategies Against Preeclampsia
Acronym: APHERESE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: INSERM UMR-S 1139 (Unknown)
Responsible Party: Sponsor
Other Study IDs: SC3455
Record Dates: First submitted 2017-04-13; First posted 2017-06-16 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; apheresis; sflt-1
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 22 Weeks
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- preeclampsia: pregnancy with preeclampsia
  Interventions: Biological: A collection of maternal plasma and serum
- control: pregnancy without preeclampsia
  Interventions: Biological: A collection of maternal plasma and serum

INTERVENTIONS:
Biological: A collection of maternal plasma and serum — A collection of maternal plasma and serum from patients with preeclampsia (PE) and normal pregnancy (NP)

SUMMARY:
The aim of the study is to setup a collection of maternal plasma and serum from patients with preeclampsia and normal pregnancy for in vitro validation of new therapeutics based on extra-corporal removal of sFlt-1

DETAILED DESCRIPTION:
A collection of maternal plasma and serum from patients with preeclampsia (PE) and normal pregnancy (NP) :

* Between 20WG and 23WG+6D : 20 patients with PE and 30 patients with NP
* Between 24WG and 27WG+6D : 20 patients with PE and 30 patients with NP
* Between 28WG and 31WG+6D : 20 patients with PE and 30 patients with NP
* Between 32WG and 35WG+6D : 20 patients with PE and 30 patients with NP
* Between 36WG and 40WG+6D : 20 patients with PE and 30 patients with NP

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 50 years old
* Singleton pregnancies between 20 and 41 weeks of gestation
* Preeclampsia
* Normal pregnancy

Exclusion Criteria:

* Age<18
* Infectious disease: HIV, HBV or HCV
* Multiple pregnancies
* Opposition of the patient

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: pregnancy with preeclampsia and without preeclampsia
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
ratio sFlt-1/PlGF | Day 0
  measurement of of sFlT-1 and PlGF

SECONDARY OUTCOMES:
Kinetics of these ratios sFlt-1/PlGF during pregnancy | until 5 month
  measurement of of sFlT-1 and PlGF at many times

CONTACTS AND LOCATIONS:
Overall Officials: Edouard Lecarpentier, MD, PhD, Study Director — Centre Hospitalier intercommunal de Créteil
Locations (1):
- Hopital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsatsaris V, Goffin F, Munaut C, Brichant JF, Pignon MR, Noel A, Schaaps JP, Cabrol D, Frankenne F, Foidart JM. Overexpression of the soluble vascular endothelial growth factor receptor in preeclamptic patients: pathophysiological consequences. J Clin Endocrinol Metab. 2003 Nov;88(11):5555-63. doi: 10.1210/jc.2003-030528. PMID 14602804
- [Background] Thadhani R, Hagmann H, Schaarschmidt W, Roth B, Cingoez T, Karumanchi SA, Wenger J, Lucchesi KJ, Tamez H, Lindner T, Fridman A, Thome U, Kribs A, Danner M, Hamacher S, Mallmann P, Stepan H, Benzing T. Removal of Soluble Fms-Like Tyrosine Kinase-1 by Dextran Sulfate Apheresis in Preeclampsia. J Am Soc Nephrol. 2016 Mar;27(3):903-13. doi: 10.1681/ASN.2015020157. Epub 2015 Sep 24. PMID 26405111
- [Background] Levine RJ, Maynard SE, Qian C, Lim KH, England LJ, Yu KF, Schisterman EF, Thadhani R, Sachs BP, Epstein FH, Sibai BM, Sukhatme VP, Karumanchi SA. Circulating angiogenic factors and the risk of preeclampsia. N Engl J Med. 2004 Feb 12;350(7):672-83. doi: 10.1056/NEJMoa031884. Epub 2004 Feb 5. PMID 14764923
- [Result] Trapiella-Alfonso L, Alexandre L, Fraichard C, Pons K, Dumas S, Huart L, Gaucher JF, Hebert-Schuster M, Guibourdenche J, Fournier T, Vidal M, Broutin I, Lecomte-Raclet L, Malaquin L, Descroix S, Tsatsaris V, Gagey-Eilstein N, Lecarpentier E. VEGF (Vascular Endothelial Growth Factor) Functionalized Magnetic Beads in a Microfluidic Device to Improve the Angiogenic Balance in Preeclampsia. Hypertension. 2019 Jul;74(1):145-153. doi: 10.1161/HYPERTENSIONAHA.118.12380. Epub 2019 May 13. PMID 31079531